CLINICAL TRIAL: NCT06566027
Title: A Comparison of the Effectiveness of Activator Versus the EF (Functional Education) Class II Standard in the Treatment of Severe Overjet in Angle Class II Division 1 Malocclusion in Vietnamese Population: A Randomized Controlled Trial
Brief Title: Activator vs the EF Class II Standard in the Treatment of Severe Overjet in Angle Class II Division 1 Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LamNguyenLe FOS-CTUMP
Record Dates: First submitted 2024-08-08; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Angle CII division 1, Activator, EF CII standard, severe OJ
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Dental Health Services

STUDY DESIGN:
Intervention Model Description: We designed the study to treat patients, randomly assigning them by lottery to receive either an activator or the EF (Functional Education) class II standard. The activator versus the EF (Functional Education) class II standard group consisted of 30 subjects (17 girls, 13 boys) and 30 subjects (12 girls, 18 boys), respectively. The changes in skeletal, dental, and soft tissue were recorded before, at 6 months of treatment. Blinding was not performed. After six months of treatment, the study's endpoint was reached and then selected those who achieved the standards for sampling at Can Tho University of Medicine and Pharmacy. The Can Tho University of Medicine and Pharmacy Ethics Council in Biomedical Research No. 23. 340.HV/PCT-H signed the study on April 12, 2023.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skeletal, dental, soft tissue index changes in Activator group (Experimental): Activator The researcher made wax impressions of the study's patients for both the activator and treatment monitoring. The researcher instructed the patients to use the activator device for 12-14 hours daily, with a minimum requirement of 12 hours. Precise ablation of the activator created plastic surfaces that guided the process of tooth eruption.
  Interventions: Other: Skeletal, dental, soft tissue index changes in Activator group
- Skeletal, dental, soft tissue index changes in EF class II standard group (Experimental): EF class II standard The researcher monitored the study children through therapy. The research used four types of EF class II standard appliances (Orthoplus, France). Patients were required to wear the EF class II standard device for at least 12 hours every day, including the entire night and at least 2 hours during the day.
  Interventions: Other: Skeletal, dental, soft tissue index changes in Activator group

INTERVENTIONS:
Other: Skeletal, dental, soft tissue index changes in Activator group — After being interviewed and provided by a doctor with two kinds of appliances (Activator and EF class II standard) for treating class II malocclusion, the patients choose their appliance. The patients were separated into two groups (30 in each). Group 1 was treated with an Activator appliance (Activator group), whereas Group 2 was treated with an EF class II standard appliance (EF line group)

SUMMARY:
Objective: The purpose of this study was to compare the clinical effectiveness of reducing severe overjet in Angle Class II division 1 malocclusion between Activator and the EF (Functional Education) class II standard in treating.

Methods: A randomized clinical trial was conducted on a total of ̉60 patients with an Angle Class II, division 1 malocclusion (ANB angle ≥ 4°, basic normal maxillary status), and an overjet of ≥ 6 mm in the developmental stage (CS1-CS3) who were eligible for the study. Thus, the sample consisted of 60 subjects (29 girls and 31 boys) with a mean age of 9.7 ± 1.31 years. The investigators designed the study to treat patients, randomly assigning them by lottery to receive either an activator or the EF (Functional Education) class II standard. The activator versus the EF (Functional Education) class II standard group consisted of 30 subjects (17 girls, 13 boys) and 30 subjects (12 girls, 18 boys), respectively. The changes in skeletal, dental, and soft tissue were recorded before, at 6 months of treatment. Blinding was not performed. After six months of treatment, the study's endpoint was reached.

DETAILED DESCRIPTION:
A randomized clinical trial was conducted on a total of ̉60 patients with an Angle Class II, division 1 malocclusion, and an overjet of ≥6 mm who were eligible for the study. Thus, the sample consisted of 60 subjects (29 girls and 31 boys) with a mean age of 9.7 ± 1.31 years. We designed the study to treat patients, randomly assigning them by lottery to receive either an activator or the EF (Functional Education) class II standard. The activator versus the EF (Functional Education) class II standard group consisted of 30 subjects (17 girls, 13 boys) and 30 subjects (12 girls, 18 boys), respectively. The changes in skeletal, dental, and soft tissue were recorded before, at 6 months of treatment. Blinding was not performed. After six months of treatment, the study's endpoint was reached and then selected those who achieved the standards for sampling at Can Tho University of Medicine and Pharmacy. The Can Tho University of Medicine and Pharmacy Ethics Council in Biomedical Research No. 23. 340.HV/PCT-H signed the study on April 12, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Vietnamese children between the ages of 7 and 12 with central incisors erupted
* Angle Class II division 1 malocclusion (ANB angle ≥ 4°, basic normal maxillary status)
* Severe overjet ≥ 6mm
* The developmental stage (CS1-CS3)
* No previous orthodontic treatment
* Agreeing to engage in the study

Exclusion Criteria:

* The young with crossbite
* Severe crowding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
To compare the clinical effectiveness of reducing severe overjet in Angle Class II division 1 malocclusion between Activator and the EF (Functional Education) class II standard in treating. | 6 months
  Every month, the research participants from both groups underwent regular re-examinations, during which they collected cephalometric radiographs for assessment at two specific time points: T0, before treatment, and T1 after 6 months of treatment. A Planmeca ProMax® 2D digital X-ray system (Planmeca, Poland) captured the cephalometric radiographs. The Dental Hospital used the licensed AudaxCeph program to accurately draw lines and perform measurements on the cephalometric images.

CONTACTS AND LOCATIONS:
Overall Officials: Lam Nguyen Le, PhD, Study Director — Can Tho University of Medicine and Pharmacy
Locations (1):
- Department of Orthodontics, Ho Chi Minh City Dental Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided